CLINICAL TRIAL: NCT05994638
Title: Polyphenol Rich Aerosol as a Support for Cancer Patients in Minimizing Side Effects After a Radiation Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AronPharma Sp. z o. o. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 08-AP-ONCOS
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-08

CONDITIONS: Oral Mucositis
Keywords: Radiotherapy; Head and neck cancer; Dysphagia; Oral Mucositis
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms; Deglutition Disorders | interventions — Aerosols; Hyaluronic Acid; Niacinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerosol for use in the oral cavity (Experimental): Group of 10 patients with head and neck cancer who have undergone radiotherapy
  Interventions: Dietary Supplement: Aerosol (Polyphenol-rich plant extracts, Hyaluronic Acid, Cetraria Islandica, Vitamin B3)

INTERVENTIONS:
Dietary Supplement: Aerosol (Polyphenol-rich plant extracts, Hyaluronic Acid, Cetraria Islandica, Vitamin B3) — Polyphenol-rich plant extracts, Hyaluronic Acid, Cetraria Islandica, Vitamin B3

SUMMARY:
The aim of the study is to demonstrate in a clinical condition the effectiveness of a preparation that is a mixture of plant extracts rich in polyphenolic compounds in the aspect of supporting cancer patients in minimizing side effects after a radiation therapy cycle.

DETAILED DESCRIPTION:
The study will be conducted on a group of 10 patients with head and neck cancer who have undergone radiation therapy and experience side effects such as discomfort/changes in the oral mucosa.The patients will receive an aerosol for oral use for a period of 1 month. Before and after the study, an assessment questionnaire related to the side effects of radiation therapy will be conducted, along with the MD Anderson Dysphagia Inventory questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Women and men, 18-75 years old
* Patients with head and neck cancer or other types of cancer after radiotherapy who suffer from oral mucositis
* Patients with dryness in mouth
* Signed informed consent.

Exclusion Criteria:

* Intake of supplements containing plant extracts, polyphenols or anthocyanins
* Participation in another clinical trial,
* Women who are pregnant, planning to become pregnant during the study or breastfeeding,
* Autoimmune disease, severe liver dysfunction, inflammatory bowel disease, tuberculosis, multiple sclerosis, AIDS, rheumatoid arthritis, organ transplantation.
* Hypersensitivity/allergy to any of the ingredient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Side effects after radiotherapy | Baseline, 1 month
  Based on a questionnaire

SECONDARY OUTCOMES:
Impact of dysphagia on quality of life | Baseline, 1 month
  Based on a MDADI questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersyteckie Centrum Stomatologiczne GUMed, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No